CLINICAL TRIAL: NCT07120932
Title: Effects of Emotional Freedom Techniques (EFT) on Pain, Cardiac Anxiety and Sleep Quality in Patients Undergoing Coronary Artery Bypass Graft Surgery: A Randomized Controlled Trial
Brief Title: Effects of Emotional Freedom Techniques on Pain, Cardiac Anxiety, and Sleep Quality in Coronary Artery Bypass Grafting
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hatice Balcı (Other)
Responsible Party: Sponsor-Investigator, Hatice Balcı, PhD, KTO Karatay University
Organization: KTO Karatay University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: EcemTEZ
Record Dates: First submitted 2025-07-16; First posted 2025-08-13 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Bypass Graft (CABG); Effects of Emotional Freedom Techniques (EFT)
Keywords: Coronary Artery Bypass Graft Surgery; Effects of Emotional Freedom Techniques (EFT); Pain Management; Anxiety; Sleep
MeSH Terms: conditions — Agnosia; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotional Freedom Techniques (EFT) (Experimental): Effects of Emotional Freedom Techniques (EFT)
  Interventions: Behavioral: Effects of Emotional Freedom Techniques (EFT)
- Control arm (No Intervention): Standard care will continue without intervention.

INTERVENTIONS:
Behavioral: Effects of Emotional Freedom Techniques (EFT) — Effects of Emotional Freedom Techniques (EFT)
  Arms: Emotional Freedom Techniques (EFT)

SUMMARY:
Objective: To determine the effect of Emotional Freedom Techniques (EFT) on pain, cardiac anxiety and sleep quality in patients undergoing Coronary Artery Bypass Graft (CABG) surgery.

Materials and Methods: The study will be conducted between 2025 and 2026 as a pretest-posttest, parallel design (1:1) randomized controlled trial. The study population will consist of patients undergoing coronary artery bypass grafting (CABG) at the Kütahya City Hospital Cardiovascular Surgery Department. The sample size was determined to be 66 patients, with 33 patients each in the experimental and control groups.

Measurement tools include a Personal Information Form, Visual Analog Scale (VAS), Cardiac Anxiety Scale, and Richard Campbell Sleep Scale. Data will be collected through one-on-one patient interviews.

The researcher has successfully completed a 3.5-hour EFT training program at the Boğaziçi Education Institute. EFT will be administered to the patients by the researcher.

Patients undergoing coronary artery bypass graft surgery at the Cardiovascular Surgery Clinic who volunteer to participate in the study and meet the inclusion criteria will complete the Informed Consent Form, Personal Information Form, Visual Analogue Scale (VAS), Cardiac Anxiety Scale, and Richard-Campbell Sleep Scale. Patients will then be assigned to the experimental or control groups by a person other than the researcher based on the randomization list. Patients in the experimental group will receive EFT in addition to standard cardiovascular surgery clinic procedures, while patients in the control group will receive standard cardiovascular surgery clinic procedures. Data analysis will be conducted using SPSS. The study will be conducted in accordance with the principles of the Declaration of Helsinki.

Findings: The findings of the research will be written after the data to be obtained after the implementation of the research and data collection will be analyzed in the SPSS program.

Conclusion: The results of the research will be written by determining the findings after analyzing the data to be obtained after the implementation of the research and data collection in the SPSS program.

ELIGIBILITY:
Inclusion Criteria: Patients who are:

* 18 years of age or older,
* 3 days postoperatively after coronary artery bypass graft surgery,
* literate,
* conscious and able to communicate will be included.

Exclusion Criteria:

* Patients with speech, hearing, or visual impairments
* Patients who do not believe in the effectiveness of the procedure due to prejudice will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
The Effect of Emotional Freedom Techniques (EFT) on Pain Levels in Patients Undergoing Coronary Artery Bypass Graft Surgery | The application, which will last 1 week for each patient, is planned for 15.09.2025-15.12.2025 dates.
  The effect of EFT on the patient's pain level will be measured. The Effect of Emotional Freedom Techniques (EFT) on Pain Levels in Patients Undergoing Coronary Artery Bypass Graft Surgery. The measurement tool is a Visual Analog Scale (VAS).

SECONDARY OUTCOMES:
The Effect of Emotional Freedom Techniques (EFT) on Cardiac Anxiety Levels in Patients Undergoing Coronary Artery Bypass Graft Surgery | The application, which will last 1 week for each patient, is planned for 15.09.2025-15.12.2025 dates.
  The effect of EFT on the patient's cardiac anxiety level will be measured. The Effect of Emotional Freedom Techniques (EFT) on Cardiac Anxiety Levels in Patients Undergoing Coronary Artery Bypass Graft Surgery. The measurement tool is a Cardiac Anxiety Scale.

OTHER OUTCOMES:
The Effect of Emotional Freedom Techniques (EFT) on Sleep Quality in Patients Undergoing Coronary Artery Bypass Graft Surgery | The application, which will last 1 week for each patient, is planned for 15.09.2025-15.12.2025 dates.
  The effect of EFT on the patient's sleep quality will be measured. The Effect of Emotional Freedom Techniques (EFT) on Sleep Quality in Patients Undergoing Coronary Artery Bypass Graft Surgery. The measurement tool is a Richard Campbell Sleep Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- KTO Karatay University, Konya, Karatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared in accordance with personal data protection laws. However, if requested by the journal boards involved in an academic publication, data will be shared within ethical limits.